CLINICAL TRIAL: NCT03935659
Title: Negative Pressure Wound Therapy for Surgical Site Infection Prevention in Vascular Surgery Patients Undergoing Common Femoral Artery Exposure
Brief Title: Negative Pressure Wound Therapy for Surgical Site Infection Prevention in Common Femoral Artery Exposure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not recruiting patients.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, loay kabbani, MD, Principle Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11956
Record Dates: First submitted 2019-04-25; First posted 2019-05-02 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Surgical Site Infection; Groin Infections
Keywords: Negative Pressure Wound Therapy
MeSH Terms: conditions — Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Patient fulfilling the inclusion criteria will be randomized into a standard gauze therapy group or a negative pressure wound therapy group.
Masking Description: As this intervention necessitated the use of an external negative wound therapy device, masking is not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard gauze therapy (Active Comparator): The control group will receive a standard sterile gauge dressing over the groin incision. The dressing will be removed on post-operative day #2 and the wound will be inspected for any complications, followed by daily dressing changes and wound inspections until discharge.
  Interventions: Procedure: Standard Wound Care
- Negative Pressure wound therapy (Experimental): The intervention group will receive a negative pressure dressing which will be applied in the operating room under sterile conditions. The brand of negative pressure dressing will be based on surgeon preference or center availability. The NPWT dressing will be removed on day 5 postoperatively or at discharge, whichever occurs first, and the groin wound inspected for any evidence of infection or dehiscence, and daily thereafter until discharge.
  Interventions: Device: Negative Pressure Pressure Wound Therapy

INTERVENTIONS:
Device: Negative Pressure Pressure Wound Therapy — Investigators will be using a Negative Pressure Wound Therapy Powered Suction Pump on primarily closed groin wounds after open common femoral artery exposure, The Negative pressure dressing will be applied in a sterile fashion in the operating room. The negative pressure dressing will be removed at day 5 postoperatively, or at discharge, whichever occurs first.
  Arms: Negative Pressure wound therapy
Procedure: Standard Wound Care — Standard sterile gauze coverage of the primarily closed groin wound.
  Arms: Standard gauze therapy

SUMMARY:
The purpose of this randomized clinical trial is to investigate the role of negative pressure wound therapy (NPWT) vs standard sterile gauze therapy on the incidence of surgical site infections (SSI) in primarily closed groin incisions in high risk patients undergoing any open common femoral artery exposure for a vascular surgery procedure.

DETAILED DESCRIPTION:
Eligible patients are randomized pre-operatively into either a standard dressing or NPWT for the groin incision.

* 1 The control group receive a standard sterile gauge dressing over the groin incision. The dressing is removed on post-operative day #2 and the wound is inspected for a SSI or dehiscence, followed by daily dressing changes and wound inspections until discharge.
* 2 The intervention group will receive a NPWT dressing which will be applied in the operating room under sterile conditions. The NPWT dressing will be removed on Post operative day 5. The wound is inspected for a SSI or dehiscence, followed by daily dressing changes and wound inspections until discharge.

ELIGIBILITY:
Inclusion Criteria: One or more of the following

* Body Mass Index >30 kg/m2
* Critical limb ischemia defined by Ankle Brachial Index<0.35, rest pain, tissue loss and/or non-healing ulcers
* Procedure time >240 min
* End Stage Renal Disease on dialysis
* Glycated hemoglobin ≥ 8.5%
* Transfusion ≥ 3 units packed Red Blood Cells
* Previous femoral artery cut-down

Exclusion Criteria:Any of the following

* Preexisting groin infection
* Complete vacuum seal cannot be achieved with negative pressure device
* Allergy to Adhesive Material
* Groin Surgery within last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Superficial surgical site infection | 30 days postoperatively
  Surgical site infection as defined by the Center for disease control and prevention criteria

SECONDARY OUTCOMES:
Mortality | 30 days
  Occurrence of mortality within 30 days of surgery
Limb Loss | 30 days and 1 year
  Occurrence of ipsilateral limb loss SSI within 30 days and 1 year of surgery
Emergency department visit for wound complication | within 30 days of surgery
  Number of participants returning to the emergency department for wound complications within 30 days of surgery
Local reaction to negative wound dressing | 5 days postoperatively
  Occurrence of a local reaction at the site of the negative pressure apparatus during application

CONTACTS AND LOCATIONS:
Overall Officials: Loay Kabbani, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cassini A, Plachouras D, Eckmanns T, Abu Sin M, Blank HP, Ducomble T, Haller S, Harder T, Klingeberg A, Sixtensson M, Velasco E, Weiss B, Kramarz P, Monnet DL, Kretzschmar ME, Suetens C. Burden of Six Healthcare-Associated Infections on European Population Health: Estimating Incidence-Based Disability-Adjusted Life Years through a Population Prevalence-Based Modelling Study. PLoS Med. 2016 Oct 18;13(10):e1002150. doi: 10.1371/journal.pmed.1002150. eCollection 2016 Oct. PMID 27755545
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1999 Apr;27(2):97-132; quiz 133-4; discussion 96. PMID 10196487
- [Background] Davis FM, Sutzko DC, Grey SF, Mansour MA, Jain KM, Nypaver TJ, Gaborek G, Henke PK. Predictors of surgical site infection after open lower extremity revascularization. J Vasc Surg. 2017 Jun;65(6):1769-1778.e3. doi: 10.1016/j.jvs.2016.11.053. PMID 28527931
- [Background] Adam DJ, Beard JD, Cleveland T, Bell J, Bradbury AW, Forbes JF, Fowkes FG, Gillepsie I, Ruckley CV, Raab G, Storkey H; BASIL trial participants. Bypass versus angioplasty in severe ischaemia of the leg (BASIL): multicentre, randomised controlled trial. Lancet. 2005 Dec 3;366(9501):1925-34. doi: 10.1016/S0140-6736(05)67704-5. PMID 16325694
- [Background] Kalish JA, Farber A, Homa K, Trinidad M, Beck A, Davies MG, Kraiss LW, Cronenwett JL; Society for Vascular Surgery Patient Safety Organization Arterial Quality Committee. Factors associated with surgical site infection after lower extremity bypass in the Society for Vascular Surgery (SVS) Vascular Quality Initiative (VQI). J Vasc Surg. 2014 Nov;60(5):1238-1246. doi: 10.1016/j.jvs.2014.05.012. Epub 2014 Jun 20. PMID 24953898
- [Background] Wiseman JT, Guzman AM, Fernandes-Taylor S, Engelbert TL, Saunders RS, Kent KC. General and vascular surgery readmissions: a systematic review. J Am Coll Surg. 2014 Sep;219(3):552-69.e2. doi: 10.1016/j.jamcollsurg.2014.05.007. Epub 2014 May 22. No abstract available. PMID 25067801
- [Background] Greenblatt DY, Rajamanickam V, Mell MW. Predictors of surgical site infection after open lower extremity revascularization. J Vasc Surg. 2011 Aug;54(2):433-9. doi: 10.1016/j.jvs.2011.01.034. Epub 2011 Mar 31. PMID 21458203
- [Background] Lee K, Murphy PB, Ingves MV, Duncan A, DeRose G, Dubois L, Forbes TL, Power A. Randomized clinical trial of negative pressure wound therapy for high-risk groin wounds in lower extremity revascularization. J Vasc Surg. 2017 Dec;66(6):1814-1819. doi: 10.1016/j.jvs.2017.06.084. Epub 2017 Aug 31. PMID 28865981
- [Background] Coomer NM, Kandilov AM. Impact of hospital-acquired conditions on financial liabilities for Medicare patients. Am J Infect Control. 2016 Nov 1;44(11):1326-1334. doi: 10.1016/j.ajic.2016.03.025. Epub 2016 May 9. PMID 27174461
- [Background] Conte MS, Bandyk DF, Clowes AW, Moneta GL, Seely L, Lorenz TJ, Namini H, Hamdan AD, Roddy SP, Belkin M, Berceli SA, DeMasi RJ, Samson RH, Berman SS; PREVENT III Investigators. Results of PREVENT III: a multicenter, randomized trial of edifoligide for the prevention of vein graft failure in lower extremity bypass surgery. J Vasc Surg. 2006 Apr;43(4):742-751; discussion 751. doi: 10.1016/j.jvs.2005.12.058. PMID 16616230
- [Background] Wiseman JT, Fernandes-Taylor S, Barnes ML, Saunders RS, Saha S, Havlena J, Rathouz PJ, Kent KC. Predictors of surgical site infection after hospital discharge in patients undergoing major vascular surgery. J Vasc Surg. 2015 Oct;62(4):1023-1031.e5. doi: 10.1016/j.jvs.2015.04.453. Epub 2015 Jul 3. PMID 26143662
- [Background] Leekha S, Lahr BD, Thompson RL, Sampathkumar P, Duncan AA, Orenstein R. Preoperative risk prediction of surgical site infection requiring hospitalization or reoperation in patients undergoing vascular surgery. J Vasc Surg. 2016 Jul;64(1):177-84. doi: 10.1016/j.jvs.2016.01.029. Epub 2016 Feb 27. PMID 26926939
- [Background] Virkkunen J, Heikkinen M, Lepantalo M, Metsanoja R, Salenius JP; Finnvasc Study Group. Diabetes as an independent risk factor for early postoperative complications in critical limb ischemia. J Vasc Surg. 2004 Oct;40(4):761-7. doi: 10.1016/j.jvs.2004.07.040. PMID 15472606
- [Background] Tan TW, Farber A, Hamburg NM, Eberhardt RT, Rybin D, Doros G, Eldrup-Jorgensen J, Goodney PP, Cronenwett JL, Kalish JA; Vascular Study Group of New England. Blood transfusion for lower extremity bypass is associated with increased wound infection and graft thrombosis. J Am Coll Surg. 2013 May;216(5):1005-1014.e2; quiz 1031-3. doi: 10.1016/j.jamcollsurg.2013.01.006. Epub 2013 Mar 25. PMID 23535163
- [Background] Semsarzadeh NN, Tadisina KK, Maddox J, Chopra K, Singh DP. Closed Incision Negative-Pressure Therapy Is Associated with Decreased Surgical-Site Infections: A Meta-Analysis. Plast Reconstr Surg. 2015 Sep;136(3):592-602. doi: 10.1097/PRS.0000000000001519. PMID 26313829
- [Background] Matatov T, Reddy KN, Doucet LD, Zhao CX, Zhang WW. Experience with a new negative pressure incision management system in prevention of groin wound infection in vascular surgery patients. J Vasc Surg. 2013 Mar;57(3):791-5. doi: 10.1016/j.jvs.2012.09.037. Epub 2013 Jan 9. PMID 23312938
- [Background] Kwon J, Staley C, McCullough M, Goss S, Arosemena M, Abai B, Salvatore D, Reiter D, DiMuzio P. A randomized clinical trial evaluating negative pressure therapy to decrease vascular groin incision complications. J Vasc Surg. 2018 Dec;68(6):1744-1752. doi: 10.1016/j.jvs.2018.05.224. Epub 2018 Aug 17. PMID 30126781
- [Background] Szilagyi DE, Smith RF, Elliott JP, Vrandecic MP. Infection in arterial reconstruction with synthetic grafts. Ann Surg. 1972 Sep;176(3):321-33. doi: 10.1097/00000658-197209000-00008. No abstract available. PMID 4262892
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585
- See also: CDC Criteria for Surgical Site Infection — https://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf